CLINICAL TRIAL: NCT00286637
Title: Novel Diagnostics for Ocular Structure
Brief Title: Novel Glaucoma Diagnostics
Status: Recruiting | Type: Observational
Sponsor: Wills Eye (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2023-37 - R01EY013178; R01EY013178 (NIH)
Record Dates: First submitted 2006-02-02; First posted 2006-02-03 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Glaucoma; Macular Disease
Keywords: OCT; CSLO; SLP; Perimetry; electrophysiology; glaucoma; macular degeneration; retinopathy; diabetes; macular hole
MeSH Terms: conditions — Glaucoma; Macular Degeneration; Retinal Diseases; Diabetes Mellitus; Retinal Perforations

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Cross-Sectional Study: Subjects will undergo a comprehensive ocular examination at every visit. Frequency of the visits is dictated by the treating physician, disregarding participation in the study. In glaucoma clinic patients are typically scheduled for visits every six months, and the frequency of visits varies according to clinical severity in the retina clinic. No additional research visits are required beyond the clinically dictated schedule.
- Longitudinal Study: Subjects will undergo a comprehensive ocular examination at every visit. Frequency of the visits is dictated by the treating physician, disregarding participation in the study. In glaucoma clinic patients are typically scheduled for visits every six months, and the frequency of visits varies according to clinical severity in the retina clinic. No additional research visits are required beyond the clinically dictated schedule.
- Reproducibility Study: Subjects willing to participate in the reproducibility arm of the project will undergo the same comprehensive ocular examination as in the longitudinal and cross-sectional study arms. However, OCT scanning will be repeated up to five times within a single visit. The participants will be requested to repeat the visual field and OCT scanning in up to 5 additional independent visits within a month to minimize the possibility that an actual change in ocular structures has occurred. Duration of each additional visit will be up to 45 minutes.
- Alzheimer's Disease (AD) Sub-Study: Participants with AD or mild cognitive impairment (MCI) undergo the same comprehensive ocular examination as in the longitudinal and cross-sectional study arms.

SUMMARY:
The purpose of this research is to evaluate novel technologies for the assessment of ocular structure and function, including the scanning device called Optical Coherence Tomography (OCT). We will test the OCT and other devices in their ability to image diseases of the eye and also compare the measurements made with OCT to those of other imaging and visual field devices approved by the Food and Drug Administration (FDA). OCT may be useful for the early diagnosis and monitoring of a variety of types of eye diseases

DETAILED DESCRIPTION:
Objective:

The purpose of this research is to evaluate a new technology, optical coherence tomography (OCT), to image diseases of the eye and to compare the measurements obtained using OCT with those of other imaging and visual field devices. OCT may be useful for the early diagnosis and monitoring of a variety of eye diseases such as age-related macular degeneration (ARMD), glaucoma, diabetic retinopathy, macular edema, and other pathologies.

Specific Aims:

There are four sub-studies: cross-sectional, longitudinal, reproducibility, and an Alzheimer's Disease (AD) sub-study. The cross-sectional and longitudinal arms study the effectiveness of the OCT technology in terms of detecting and monitoring eye diseases. The reproducibility study is designed to test the measurement likeness of the OCT. The AD sub-study will use high resolution ocular imaging technologies to determine ocular biomarkers for sensitive detection of AD.

Background:

This is a continuation of an ongoing study from the New England Eye Center (NEEC), Tufts Medical Center, Boston, MA. This study started when our research group was located at NEEC and in collaboration with the Massachusetts Institute of Technology (MIT) where we conducted the first clinical studies with OCT. The first investigation using OCT was published in Science in 1991 and showed in vitro imaging of the human retina and atherosclerotic plaque. We developed an OCT prototype system for performing preliminary ophthalmic clinical studies and in 1993, began clinical OCT imaging studies.

The prototype ophthalmic OCT instrument acquired OCT images of the retina with an axial resolution of 10µm within an acquisition time of 2.5 sec. The OCT imaging system was integrated with a slit-lamp biomicroscope for in vivo tomography of the anterior and posterior eye. The beam is directed into the eye using computer controlled galvonometric scanners, which can scan arbitrary transverse patterns. The beam focus is coincident with the slit-lamp image plane to permit simultaneous scanning and visualization of the eye through the slit-lamp or via a CCD camera. For tomography of the anterior eye, the microscope is focused directly on the structure, while for retinal imaging, a lens relay images of the retina onto the slit-lamp image plane. A computer provides real-time display of the tomogram, image processing, and data management.

OCT technology was patented and subsequently transferred to industry (Zeiss Humphrey Systems, CA). Our prototype ophthalmic OCT system was developed into a clinical instrument and was introduced into the ophthalmic market in 1996. The commercial OCT technology has an axial resolution of 10 µm and can acquire a 100 transverse pixel retinal tomogram in 1 second. A third generation ophthalmic OCT imaging device, OCT3, was introduced three years ago. OCT imaging is now used as a standard diagnostic procedure as part of an ophthalmic examination for many retina and glaucoma patients at the University of Pittsburgh Medical Center (UPMC) Eye Center and New England Eye Center (NEEC). OCT imaging is in use in major research and clinical centers internationally. The OCT has been approved by the Food and Drug Administration for use in ophthalmology.

Significance:

OCT enables tissue pathology to be imaged in situ and in real time with a resolution approaching that of conventional histopathology but without the need for excising and processing specimens. OCT provides a quantitative method of directly measuring ocular structures with high precision and could provide an objective, early diagnosis for glaucoma, age related macular degeneration (ARMD), diabetic retinopathy, macular edema, and other pathologies. Extensive studies have been performed with OCT in cross-sectional as well as longitudinal setting. In this ongoing protocol, our objective is to continue these studies using the commercial ophthalmic OCT imaging instruments to develop methods for early detection and improve longitudinal assessment for the above mentioned ocular pathologies.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent and to understand the study procedures
* Healthy volunteers
* Age related macular degeneration (AMD), diabetic retinopathy, central serous chorioretinopathy, and/or glaucoma or glaucoma suspects
* (AD Sub-Study ONLY): Subjects diagnosed with AD or MCI.

Exclusion Criteria:

* Any medical treatment (e.g., chronic corticosteroid, hydroxychloroquine, chloroquine, thioridazine, canthaxanthine) or conditions that affect VF (e.g., stroke) and retinal thickness other than glaucoma.
* Strabismus, nystagmus, or any condition that prevents fixation.
* Presence of any media opacities that hinders clinical view of the fundus, and any intraocular non-glaucomatous abnormality
* History of ocular trauma or intraocular surgery other than uncomplicated glaucoma interventions or cataract extraction at least 3 months previous to participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study aims to enroll healthy volunteers and subjects with glaucoma, age related macular degeneration (AMD), diabetic retinopathy (DR), and central serous chorioretinopathy (CSCR). Participants with AD and MCI will be recruited as part of a sub-study.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2000-08-01 (Actual); Primary Completion 2029-07-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants who Show Evidence of Glaucoma Progression | Up to Year 5
  The purpose of this research is to Participants who show evidence of glaucoma progression are classified as "progressors." Participants who show evidence of glaucoma progression are classified as "progressors."

CONTACTS AND LOCATIONS:
Overall Officials: Joel S Schumann, MD, Study Chair — Wills Eye Hospital
Locations (1):
- Wills Eye Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mumcuoglu T, Townsend KA, Wollstein G, Ishikawa H, Bilonick RA, Sung KR, Kagemann L, Schuman JS; Advanced Imaging in Glaucoma Study Group. Assessing the relationship between central corneal thickness and retinal nerve fiber layer thickness in healthy subjects. Am J Ophthalmol. 2008 Oct;146(4):561-6. doi: 10.1016/j.ajo.2008.05.038. Epub 2008 Jul 26. PMID 18657796
- [Derived] Gabriele ML, Ishikawa H, Wollstein G, Bilonick RA, Townsend KA, Kagemann L, Wojtkowski M, Srinivasan VJ, Fujimoto JG, Duker JS, Schuman JS. Optical coherence tomography scan circle location and mean retinal nerve fiber layer measurement variability. Invest Ophthalmol Vis Sci. 2008 Jun;49(6):2315-21. doi: 10.1167/iovs.07-0873. PMID 18515577